CLINICAL TRIAL: NCT02755662
Title: Clinical Impact of 2 Types of Mandibular Retention Devices - Narval O.R.M Cad Cam Design vs Narval O.R.M Traditional Design - on Obstructive Sleep Apnea Syndrome (OSA) Therapy: ESTAMPS Study
Brief Title: Clinical Impact of 2 Types of Mandibular Retention Devices - Narval O.R.M CadCam Design vs Narval O.R.M Traditional Design - on Obstructive Sleep Apnea (OSA) Therapy: ESTAMPS Study
Acronym: ESTAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RESMED Estamps 001
Record Dates: First submitted 2016-04-07; First posted 2016-04-29 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; mandibular repositioning device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narval O.R.M CC™ (Active Comparator): First mandibular retention device : Narval O.R.M CC™
  Interventions: Device: Mandibular Retention Device
- Narval O.R.M™ trad (Active Comparator): Second mandibular retention device : Narval O.R.M TRAD™
  Interventions: Device: Mandibular Retention Device

INTERVENTIONS:
Device: Mandibular Retention Device
  Other Names: Narval O.R.M CC™

SUMMARY:
ESTAMPS is a randomized clinical trial with a crossover design:

Main objective is to compare impact of 2 different Mandibular Retention Device (MRD) designs (Narval MRD CadCam (CC) design vs Narval MRD traditional (trad) design) on upper airway volume

secondary objectives: To evaluate the maximal mandibular propulsion according to the type of MRD To evaluate benefits on quality of life, sleepiness and OSA symptoms To evaluate impact of MRD design on therapy efficacy and tolerance To evaluate impact of MRD design on mandibular positioning

DETAILED DESCRIPTION:
Hypothesis ORCADES results suggest that Narval O.R.M CC could be more efficient than Narval MRD trad to reduce AHI whatever the initial OSA severity 79% of CC MRD patients have at least an AHI reduction of 50% (vs. 61% with a trad Narval MRD, p=0.0031) 66% of CC MRD patients get a complete answer with an AHI reduction <10 (vs. 49% with a trad Narval MRD, p=0.0017) The investigators think that differences seen in the ORCADES study between the 2 MRD is due to a different impact on upper airway volume

ELIGIBILITY:
Inclusion Criteria:

* Patients with a mild OSA syndrome (5<AHI<30) and mild to moderate sleepiness without cardiac comorbidities or patients with mild to severe OSA syndrome (IAH>15) who do not tolerate or refuse CPAP therapy
* Patients ≥ 18 years old
* Patient is able to fully understand study information and provide written informed consent

Exclusion Criteria:

* MRD contraindication
* Clinical trial classic exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
upper airway volume | 1 month
  investigators will measure upper airway volume (cm3) changes produced by 2 different Mandibular Retention Devices in Obstructive sleep apnea syndrome (OSA) patients

SECONDARY OUTCOMES:
maximal mandibular propulsion | 1 month
  investigators will measure the maximal mandibular propulsion (in millimeter) at the end of MRD titration
quality of sleep | 1 month
  investigators will use specific quality of sleep questionnaire: Pittsburgh sleep quality index (PSQI),
sleepiness | 1 month
  investigators will use a specific sleepiness questionnaire: Epworth sleepiness scale (ESS)
MRD therapy efficacy | 1 month
  investigators will measure the residual Apnea and Hypopnea Index (AHI) via polygraphy
mandibular positioning | 1 month
  investigators will measure the mandibular positioning under MRD therapy (in millimeter)
Occlusal vertical dimension | 1 month
  investigators will measure the occlusal vertical dimension changes (in millimeter) between the 2 type of MRD

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Kerbrat, MD, Principal Investigator — CHU Rouen
Locations (1):
- CHU Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No